CLINICAL TRIAL: NCT06143540
Title: Clinical Study of 18F Labeled Probe Targeting Fibroblast Activating Protein and Integrin avβ3 (FAPI-RGD) in Interstitial Lung Disease Associated With Connective Tissue Disease
Brief Title: Clinical Study of 18F-FAPI-RGD in Interstitial Lung Disease Associated With Connective Tissue Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Other Study IDs: SCPH-ILDCTD
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine clinical utility of 18F-FAPI-RGD PET/CT imaging in evaluating connective tissue disease-associated interstitial lung disease. Participants will undergo clinical evaluation and 18F-FAPI-RGD PET/CT examination.

DETAILED DESCRIPTION:
Interstitial lung disease is an overarching term for a wide range of disorders characterized by inflammation and/ or fibrosis in the lungs. Interstitial lung disease associated connective tissue diseases(CTD-ILD) is one of the most common types.The goal of this study is to explore the feasibility of using 18F-FAPI-RGD, a dual-targeting heterodimeric PET tracer that recognizes both fibroblast activation protein (FAP) and integrin αvβ3 for detecting connective tissue disease associated interstitial lung disease (CTD-ILD), and analyze the relationship between 18F- FAPI-RGD PET/CT images and related parameters of lung function, clinical laboratory indicators and HRCT scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients who have been diagnosed with, or are clinically highly suspected of ILD
* Patients who have been diagnosed with, or are clinically highly suspected of CTD-ILD

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients with tumor, other respiratory diseases, and lung surgery
* Abnormal cardiopulmonary function or mental state, unable tolerate PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or diagnosed connective tissue disease-associated interstitial lung disease
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical indicators and PET/CT results | 2 months
  Correlation of clinical pulmonary function indexes, HRCT, laboratory examination indexes and 18F-FAPI-RGD PET/CT results

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China